CLINICAL TRIAL: NCT03866070
Title: Efficacy of a Physiotherapy Intervention by Stretching the Posterior Capsule of the Shoulder in the Stability of the Glenohumeral Joint and the Throwing Performance in Handball Players. A Randomized Clinical Trial
Brief Title: Stretching the Posterior Capsule of the Shoulder in the Stability and the Throwing Performance in Handball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ECEF
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Shoulder Injuries and Disorders
Keywords: Handball; Physiotherapy; Shoulder instability; Scapular dyskinesia; Female
MeSH Terms: conditions — Shoulder Injuries; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The subjects that are part of the experimental group will carry out the intervention thought the performance of strengthening exercises of the shoulder and scapula, and capsular stretches.
  Interventions: Other: Experimental
- Control (Active Comparator): Subjects that are part of the control group will perform shoulder strengthening exercises exclusively.
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — Two exercises will be done to strengthen the external rotation (using elastic bands): standing with 90 degrees of shoulder abduction and elbow flexion and also in standing with the shoulder in neutral position and the elbow flexed to 90 degrees. Subjects will perform 3 sets of 10 repetitions with the band slightly stretched, at a distance of 0.70 m from the wall. Dumbbell exercises will be performed through 4 exercises: flexion in the horizontal plane of 135º, external rotation in lateral decubitus, horizontal abduction with external rotation, and extension in prone position. There will be 5 repetitions each exercise of 3 seconds each, with 2 minutes of rest between exercises.
  Other Names: Strengthening exercises and capsular stretches
  Arms: Experimental
Other: Control — Two exercises will be done to strengthen the external rotation, using elastic bands. The first, standing, with 90 degrees of shoulder abduction and elbow flexion. The second, also in standing, with the shoulder in neutral position and the elbow flexed to 90 degrees. Subjects will perform 3 sets of 10 repetitions with the band slightly stretched, at a distance of 0.70 m from the wall. The band will be subject to a surface, at an equal distance from the subject's elbow to the ground. The repetitions will last one second in concentric external rotation and two seconds in eccentric external rotation, with a rest of 30 seconds between series.
  Other Names: Strengthening exercises
  Arms: Control

SUMMARY:
Introduction: Handball is a sport with a high prevalence of shoulder injuries due to the overuse that causes a glenohumeral internal rotation deficit, and excess of external rotation and scapular dyskinesia. Stretching is essential to restore physiological movement and improve strength.

Aim: To evaluate the efficacy of a posterior capsule stretching and strengthening of the shoulder and scapular program in handball players from 18 to 37 years old.

Study design: randomized clinical trial, multicenter, single-blind with follow-up period.

Methods: 60 handball players will be randomly assigned to the two study groups (experimental and control). The intervention will last 4 weeks, with 3 weekly sessions with a duration of 21 and 12 minutes each. The study variables will be: range of motion in internal and external rotation (goniometer), throwing speed (Ball Throwing Speed Test), functionality (DASH questionnaire), perceived exertion (Borg scale), glenohumeral stability (CKCUEST y YBT-UQ Test) and the throwing force (Overhead Medicine Ball Throw). The intervention will consist in the application of stretching of the posterior shoulder capsule with an exercise protocol. A Kolmogorov-Smirnov analysis will calculate the normality of the distribution. In case of homogeneity of the groups, with the t-student test of repeated measurements and an ANOVA of repeated averages, the difference between the different evaluations and the intra- and inter-subject effect will be calculated.

Expected results: Improved range of motion of the shoulder, strength and throwing speed after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Handball players federated in the Madrid Handball Federation
* With an age range between 18 and 37 years
* More than 2 years of handball sports
* Currently participate in amateur competitions of First National Women's category.

Exclusion Criteria:

* Have suffered a shoulder injury in the last six months
* Who are currently doing some physiotherapy treatment
* Who fail to participate in the established intervention and evaluation sessions
* Refusing to sign the informed consent document.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline functionality of the shoulder after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The functionality of the shoulder will be measured with the questionnaire Disability of the Arm, Shoulder and Hand (DASH). This scale consists of 30 items (of functionality). The score range of this scale ranges from 0 to 100 points (where a higher score indicates less functionality).

SECONDARY OUTCOMES:
Change from baseline perception of effort after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The perception of effort will be measured with the modified Borg scale. In this instrument, 11 items are evaluated, with a score of 0 to 10 points, where 0 equals the minimum effort and 10 the maximum that they can perform.
Change from baseline launch speed after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The launch speed with the handball (56 cm and 375 grams of weight) will be measured using the Ball Throwing Speed Test. This measuring instrument requires the use of a stopwatch. The measurement will be made through the execution of 6 launches. The athletes must have both feet resting on the ground at a distance of 2.5 meters from the wall, making the throws at maximum speed, collecting the best result. The unit of measurement of this test is meters / second (where the higher the score, the faster the launch).
Change from baseline shoulder stability after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The assessment of shoulder stability will be carried out using the Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST). The player will be placed in the ironing position with the arms extended and supported on the ground. The objective is to assess how many times it is able to raise the arm to touch the opposite shoulder in 15 seconds. This test is measured by the number of repetitions you perform (the greater the number of repetitions, the better the stability of the shoulder).
Change from baseline distance range after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Distance range will be calculated using the Upper Quarter Y-Balance Test (YBT-UQ Test). We will use 3 different angles from where the handball players, with a support arm, should push an object on a tape measure. This test measures the stability and mobility of the upper limbs of the body. The unit of measurement for this test is centimeters (the greater the distance traveled in cm, the better the reach distance of the upper limbs).
Change from baseline strength of upper limbs after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The strength of upper limbs will be evaluated with Overhead Medicine Ball Throw (OMBT). The athletes, with both feet resting on the ground and using a reference point "0" of the tape measure, will throw a medicine ball over the head in order to reach the greatest possible distance. This distance will be measured with a tape measure, the meter being the unit of measurement the centimeter (the greater the distance, the greater the strength of the upper limbs)
Change from baseline shoulder range of motion after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The measurement of the range of movement of the shoulder will be made with a universal goniometer. The movements of external and internal rotation will be measured. The women will be in the supine position with the scapula and the spine stabilized. The goniometer axis will be placed in the olecranon, while the fixed arm will be located vertical to the axis of the humerus, and the mobile arm parallel to the forearm by the ulna axis. The unit of measurement will be in degrees, with the normal range of mobility being 70 to 90 degrees in internal and external rotation, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain